CLINICAL TRIAL: NCT02152800
Title: A Study of Vacyless® Versus Valtrex® in Patients With Herpes Zoster
Acronym: Vacyless®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RCH3002P02
Record Dates: First submitted 2014-03-13; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vacyless® 1000 mg (Experimental): one Vacyless® 1000 mg tablets, 3 times daily for 7days
  Interventions: Drug: valacyclovir hydrocholoride
- Vacyless® 500mg (Experimental): Two Vacyless® 500mg tablets, 3 times daily for 7 days
  Interventions: Drug: valacyclovir hydrocholoride
- Valtrex® 500 mg (Active Comparator): Two Valtrex® 500 mg tablets, 3 times daily for 7days
  Interventions: Drug: valacyclovir hydrocholoride

INTERVENTIONS:
Drug: valacyclovir hydrocholoride

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Vacyless® and Valtrex® in patients with acute herpes zoster.

DETAILED DESCRIPTION:
Primary Endpoint:

- Lesion assessment - Rash severity, in terms of rash counts

Secondary Endpoints:

* Pain assessment
* Clinical global impression
* Safety information of valacyclovir

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 to 80 years of age.
* Patients with a clinical diagnosis of HZ as evidenced by a unilateral dermatomal rash.
* Patients with zoster-related rash (rash severity is greater than or equal to mild).
* Patients are able to be enrolled into the study 72 hours from appearance of rash (for example, lesions or vesicles).
* Patients provided written informed consent.
* Patients who are able to complete all study visits per protocol.
* Men and premenopausal women must agree to practice a barrier method of birth control or the use of a spermicide for one month after the last dose of study drug (oral contraceptives are not permitted). Subject should be withdrew from the study if contraceptions are faild.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients with multidermatomal or disseminated HZ (greater than 20 lesions beyond the dermatomes adjacent to the primarily involved dermatome).
* Patients with HZ ophthalmicus, defined as cutaneous lesions in the dermatome associated with the ophthalmic division of the trigeminal nerve
* Patients with history of impaired renal function, (e.g., calculated creatinine clearance less than 50 mL/min/1.73 m2)
* Patients are taking narcotic analgesic routinely for a chronic pain condition
* Patients are taking tricyclic antidepressants
* Patients who received systemic antivirals with activity against VZV within the past 30 days, or a topical antiviral to treat their current HZ
* Patients with immunosuppressive or immunodeficient condition resulting from:

disease (e.g., HIV) corticosteroid use (except intermittent or topical/inhaled beclomethasone dipropionate or equivalent < 800 mcg/day), or other immunosuppressive/cytotoxic therapy (cancer chemotherapy or organ transplantation )

* Patients with any other condition (e.g., extensive psoriasis, chronic pain syndrome, cognitive impairment) that, in the opinion of the site investigator, might interfere with the evaluations required by the study
* Patients who are not ambulatory (bed-ridden or homebound); hospitalized patients may be enrolled if they are ambulatory and able to complete the study requirements
* Patients with history of allergy to valacyclovir hydrochloride and acetaminophen
* Patients are unlikely to adhere to protocol follow-up

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the rash severity, in terms of rash counts | Day 28

SECONDARY OUTCOMES:
VAS Pain score | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Yuan Shi, M.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan